CLINICAL TRIAL: NCT01968707
Title: Assessment of the Antimicrobial Efficacy of 3M CHG/IPA Preoperative Skin Preparation Against Resident Human Skin Flora on the Abdominal and Inguinal Regions
Brief Title: In-vivo Efficacy Study of Patient Pre-operative Preps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EM-012760
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Bacterial Reduction on Skin Flora Post-product Application
Keywords: surgical prep; CHG; IPA
MeSH Terms: interventions — chlorhexidine gluconate; Ethanol; 2-Propanol; Chromogranins; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- ChloraPrep Hi-Lite Orange (Active Comparator): Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: ChloraPrep Hi-Lite Orange
- Normal Saline (Placebo Comparator): Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: Normal saline
- 3M CHG/IPA Prep Tint 10.5 mL (Experimental): Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: 3M CHG/IPA Prep Tint 10.5-mL
- 3M CHG/IPA Prep Tint 26-mL (Experimental): Apply topically for 30 seconds to the abdominal region or 2 minutes to the inguinal region, and allow to dry for 3 minutes.
  Interventions: Drug: 3M CHG/IPA Prep Tint 26-mL

INTERVENTIONS:
Drug: ChloraPrep Hi-Lite Orange — Apply topically.
  Other Names: ChloraPrep One-Step; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%; Chlorhexidine gluconate 2% w/v / Isopropyl alcohol 70% v/v; 2% CHG / 70% IPA; ChloraPrep; Chlorhexidine Gluconate and Isopropyl alcohol
  Arms: ChloraPrep Hi-Lite Orange
Drug: Normal saline — Apply topically.
  Other Names: 0.9% Sodium Chloride; Sterile Saline; 0.9% NaCl; Saline
  Arms: Normal Saline
Drug: 3M CHG/IPA Prep Tint 10.5-mL — Apply topically.
  Other Names: Chlorhexidine Gluconate and Isopropyl Alcohol; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%; Chlorhexidine gluconate 2% w/v / Isopropyl alcohol 70% v/v; 2% CHG / 70% IPA
  Arms: 3M CHG/IPA Prep Tint 10.5 mL
Drug: 3M CHG/IPA Prep Tint 26-mL — Apply topically
  Other Names: Chlorhexidine Gluconate and Isopropyl Alcohol; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%; Chlorhexidine gluconate 2% w/v / Isopropyl alcohol 70% v/v; 2% CHG / 70% IPA
  Arms: 3M CHG/IPA Prep Tint 26-mL

SUMMARY:
The purpose of this study is to determine the antimicrobial efficacy of the 3M CHG/IPA Prep on skin flora of the abdominal and inguinal regions of human subjects.

DETAILED DESCRIPTION:
The primary efficacy is evaluated by demonstration that the product provides a lower bound of the 95% confidence interval of percent responders that is greater than or equal to 70%.

On the abdominal sites, a responder is defined as a subject with a 2-log10 per cm2 bacterial reduction at 10 minutes and for whom the skin flora does not return to baseline at 6 hours.

On the inguinal sites, a responder is defined as a subject with a 3-log10 per cm2 bacterial reduction at 10 minutes and for whom the skin flora does not return to baseline at 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any race
* Subjects in good general health
* Minimum skin flora baseline requirements on abdomen and groin

Exclusion Criteria:

* Any tattoos, scars, breaks in the skin, or any form of dermatitis, or other skin disorders (including acne) on the applicable test areas
* Topical antimicrobial exposure within 14 days prior to screening and treatment days
* Use of systemic or topical antibiotics, steroid medications, or any other products known to affect the normal microbial flora of the skin within 14 days prior to screening and treatment days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad H Bashir, MD, CCRP, Principal Investigator — MICROBIOTEST
Locations (1):
- Microbiotest, Sterling, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a randomized, paired comparison design where each subject received 2 of the planned treatments, 1 on the left side & 1 on the right. Each subject provided 2 abdomen test sites, left & right and/or 2 inguen test sites, left & right.
  406 subjects were randomized for the abdomen region & 391 subjects randomized for the inguen region resulting in 426 subjects providing 1594 applications of test products on 2 anatomical regions.
Units Other Than Participants: test sites on skin
Groups:
- ChloraPrep Hi-Lite Orange - Abdominal; Normal Saline - Abdominal; 3M CHG/IPA Prep Tint 10.5-mL - Abdominal; 3M CHG/IPA Prep Tint 26-mL - Abdominal: Applied topically to the abdominal region for 30 seconds.
- ChloraPrep Hi-Lite Orange - Inguinal; Normal Saline - Inguinal; 3M CHG/IPA Prep Tint 10.5-mL - Inguinal; 3M CHG/IPA Prep Tint 26-mL - Inguinal: Applied topically to the inguinal region for 2 minutes.
Period: Overall Study
Arm/Group | ChloraPrep Hi-Lite Orange - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep Tint 10.5-mL - Abdominal | 3M CHG/IPA Prep Tint 26-mL - Abdominal | ChloraPrep Hi-Lite Orange - Inguinal | Normal Saline - Inguinal | 3M CHG/IPA Prep Tint 10.5-mL - Inguinal | 3M CHG/IPA Prep Tint 26-mL - Inguinal
Started | 247; 247 test sites on skin | 74; 74 test sites on skin | 246; 246 test sites on skin | 245; 245 test sites on skin | 236; 236 test sites on skin | 70; 70 test sites on skin | 238; 238 test sites on skin | 238; 238 test sites on skin
Completed | 198; 198 test sites on skin | 62; 62 test sites on skin | 205; 205 test sites on skin | 201; 201 test sites on skin | 200; 200 test sites on skin | 59; 59 test sites on skin | 204; 204 test sites on skin | 203; 203 test sites on skin
Not Completed | 49; 49 test sites on skin | 12; 12 test sites on skin | 41; 41 test sites on skin | 44; 44 test sites on skin | 36; 36 test sites on skin | 11; 11 test sites on skin | 34; 34 test sites on skin | 35; 35 test sites on skin
Not completed — Did not meet treatment day baseline | 49 | 12 | 41 | 44 | 36 | 11 | 34 | 35

BASELINE CHARACTERISTICS:
Population: Subjects with average treatment day baseline counts of greater than or equal to 3.00 log10 CFU/cm2 bilaterally on the abdominal region and/or greater than or equal to 5.00 log10 CFU/cm2 bilaterally on the inguinal region were included in the analysis.
Units Other Than Participants: Test sites on skin
Groups:
- ChloraPrep Hi-Lite Orange - Abdominal: ChloraPrep 2% CHG/70% IPA 26-mL applicator applied topically for 30 seconds.
- Normal Saline - Abdominal: Normal Saline with applicator applied topically for 30 seconds.
- 3M CHG/IPA Prep Tint 10.5-mL - Abdominal: 3M CHG/IPA 2% CHG/70% IPA 10.5-mL applicator applied topically for 30 seconds.
- 3M CHG/IPA Prep Tint 26-mL - Abdominal: 3M CHG/IPA 2% CHG/70% IPA 26-mL applicator applied topically for 30 seconds.
- ChloraPrep Hi-Lite Orange - Inguinal: ChloraPrep 2% CHG/70% IPA 26-mL applicator applied topically for 2 minutes.
- Normal Saline - Inguinal: Normal Saline with applicator applied topically for 2 minutes.
- 3M CHG/IPA Prep Tint 10.5-mL - Inguinal: 3M CHG/IPA 2% CHG/70% IPA 10.5-mL applicator applied topically for 2 minutes.
- 3M CHG/IPA Prep 26-mL - Inguinal: 3M CHG/IPA 2% CHG/70% IPA 26-mL applicator applied topically for 2 minutes.
- Total: Total of all reporting groups
Arm/Group | ChloraPrep Hi-Lite Orange - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep Tint 10.5-mL - Abdominal | 3M CHG/IPA Prep Tint 26-mL - Abdominal | ChloraPrep Hi-Lite Orange - Inguinal | Normal Saline - Inguinal | 3M CHG/IPA Prep Tint 10.5-mL - Inguinal | 3M CHG/IPA Prep 26-mL - Inguinal | Total
Number analyzed (Participants) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 426
Number analyzed (Test sites on skin) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 1594
Age, Customized [Number; unit: participants]
  <=18 years | 247 | 74 | 246 | 246 | 236 | 70 | 238 | 238 | 0
  Between 18 and 65 years | 247 | 74 | 246 | 246 | 236 | 70 | 238 | 238 | 409
  >=65 years | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 17
Sex/Gender, Customized [Number; unit: participants]
  Female | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 213
  Male | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 213
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 2
  Asian | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 136
  Black or African American | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 70
  Hispanic/Latino | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 49
  Native Hawiian or Other Pacific Islander | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 2
  White | 247 | 74 | 246 | 245 | 236 | 70 | 237 | 238 | 160
  Other | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 7
Region of Enrollment [Number; unit: participants]
  United States | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238 | 426

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate
Description: On the abdominal region a responder was a subject with a 2 log10/cm2 bacterial reduction at 10 minutes and for whom the skin flora did not return to baseline.
  On the inguinal region a responder was a subject with a 3 log10/cm2 bacterial reduction at 10 minutes and for whom the skin flora did not return to baseline.
Time Frame: baseline, 10 minutes post-product application and 6 hour post-product application
Population: The primary analysis data set used a Modified Intent to Treat population. Subjects were excluded who did not meet the treatment day baseline requirements of either > or equal to 3.0 log10 on the abdomen test site or 5.0 log10 on the inguinal test site.
Measure: Count of Participants; unit: Participants
Groups:
- Normal Saline - Abdominal: Apply topically to the abdominal region for 30 seconds
- Normal Saline - Inguinal: Apply topically to the inguinal region for 2 minutes
Arm/Group | ChloraPrep Hi-Lite Orange - Abdominal | 3M CHG/IPA Prep Tint 10.5-mL - Abdominal | 3M CHG/IPA Prep Tint 26-mL - Abdominal | Normal Saline - Abdominal | ChloraPrep Hi-Lite Orange - Inguinal | 3M CHG/IPA Prep Tint 10.5-mL - Inguinal | 3M CHG/IPA Prep Tint 26-mL - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 198 | 205 | 201 | 62 | 200 | 204 | 203 | 59
Participants | 178 | 167 | 175 | 0 | 168 | 168 | 162 | 4

2. Secondary Outcome: Reduction of Skin Flora 6 Hours Post-treatment
Description: log10/cm2 reduction of skin flora, relative to treatment day baseline (log10/cm2), at 6 hours post-treatment
Time Frame: 6 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10/cm2
Arm/Group | ChloraPrep Hi-Lite Orange - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep Tint 10.5-mL - Abdominal | 3M CHG/IPA Prep Tint 26-mL - Abdominal | ChloraPrep Hi-Lite Orange - Inguinal | Normal Saline - Inguinal | 3M CHG/IPA Prep Tint 10.5-mL - Inguinal | 3M CHG/IPA Prep Tint 26-mL - Inguinal
Number analyzed (Participants) | 198 | 62 | 205 | 201 | 200 | 59 | 204 | 203
log10/cm2 | 1.77 (0.899) | 0.47 (0.651) | 1.48 (0.866) | 1.64 (0.864) | 2.64 (1.047) | 1.08 (0.833) | 2.24 (1.103) | 2.35 (1.045)

3. Secondary Outcome: Reduction of Skin Flora 10 Minutes Post-treatment
Description: log10/cm2 reduction of skin flora, relative to treatment day baseline (log10/cm2), at 10 minutes post-treatment
Time Frame: 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10/cm2
Arm/Group | ChloraPrep Hi-Lite Orange - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep Tint 10.5-mL - Abdominal | 3M CHG/IPA Prep Tint 26-mL - Abdominal | ChloraPrep Hi-Lite Orange - Inguinal | Normal Saline - Inguinal | 3M CHG/IPA Prep Tint 10.5-mL - Inguinal | 3M CHG/IPA Prep Tint 26-mL - Inguinal
Number analyzed (Participants) | 198 | 62 | 205 | 201 | 200 | 59 | 204 | 203
log10/cm2 | 2.79 (0.565) | 0.64 (0.488) | 2.66 (0.706) | 2.74 (0.644) | 4.04 (0.964) | 1.34 (1.096) | 3.98 (1.034) | 3.89 (0.929)

4. Secondary Outcome: Skin Flora Recovery 6-hours Post-treatment
Description: Log10/cm2 recovery of skin flora at 6 hours following application of study treatment
Time Frame: 6 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10/cm2 skin flora
Groups:
- ChloraPrep Hi-Lite Orange - Abdominal: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 26-mL applied topically to the abdominal region for 30 seconds.
  ChloraPrep Hi-Lite Orange Tint: Apply topically.
- Normal Saline - Abdominal: 0.9% normal saline applied topically to the abdominal region for 30 seconds.
  Normal Saline: Apply topically.
- 3M CHG/IPA Prep Tint 10.5-mL - Abdominal: Chlorhexidine gluconate 2% / Isopropyl alcohol 70% 10.5 mL applied topically to the abdominal region for 30 seconds.
  3M CHG/IPA Prep Tint 10.5-mL: Apply topically.
- 3M CHG/IPA Prep Tint 26-mL - Abdominal: Chlorhexidine gluconate 2% / Isopropyl alcohol 70% 26 mL applied topically to the abdominal region for 30 seconds.
  3M CHG/IPA Prep Tint 26-mL: Apply topically
- ChloraPrep Hi-Lite Orange - Inguinal: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 26-mL applied topically to the inguinal region for 2 minutes.
  ChloraPrep Hi-Lite Orange Tint: Apply topically.
- Normal Saline - Inguinal: 0.9% normal saline applied topically to the inguinal region for 2 minutes.
  Normal Saline: Apply topically.
- 3M CHG/IPA Prep Tint 10.5-mL - Inguinal: Chlorhexidine gluconate 2% / Isopropyl alcohol 70% 10.5 mL applied topically to the inguinal region for 2 minutes.
  3M CHG/IPA Prep Tint 10.5-mL: Apply topically.
- 3M CHG/IPA Prep Tint 26-mL - Inguinal: Chlorhexidine gluconate 2% / Isopropyl alcohol 70% 26 mL applied topically to the inguinal region for 2 minutes
  3M CHG/IPA Prep Tint 26-mL: Apply topically
Arm/Group | ChloraPrep Hi-Lite Orange - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep Tint 10.5-mL - Abdominal | 3M CHG/IPA Prep Tint 26-mL - Abdominal | ChloraPrep Hi-Lite Orange - Inguinal | Normal Saline - Inguinal | 3M CHG/IPA Prep Tint 10.5-mL - Inguinal | 3M CHG/IPA Prep Tint 26-mL - Inguinal
Number analyzed (Participants) | 198 | 62 | 205 | 201 | 200 | 59 | 204 | 203
log10/cm2 skin flora | 1.54 (0.808) | 2.80 (0.726) | 1.87 (0.804) | 1.66 (0.803) | 2.81 (1.008) | 4.31 (0.941) | 3.20 (1.037) | 3.07 (1.032)

5. Secondary Outcome: Skin Flora Recovery 10 Minutes Post-treatment
Description: Log10/cm2 recovery of skin flora at 10 minutes following application of study treatments
Time Frame: 10 minutes post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10/cm2 skin flora
Arm/Group | ChloraPrep Hi-Lite Orange - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep Tint 10.5-mL - Abdominal | 3M CHG/IPA Prep Tint 26-mL - Abdominal | ChloraPrep Hi-Lite Orange - Inguinal | Normal Saline - Inguinal | 3M CHG/IPA Prep Tint 10.5-mL - Inguinal | 3M CHG/IPA Prep Tint 26-mL - Inguinal
Number analyzed (Participants) | 198 | 62 | 205 | 201 | 200 | 59 | 204 | 203
log10/cm2 skin flora | 0.52 (0.500) | 2.63 (0.582) | 0.69 (0.604) | 0.57 (0.575) | 1.41 (1.089) | 4.06 (1.211) | 1.47 (1.120) | 1.53 (1.039)

6. Secondary Outcome: Skin Flora Baseline for the Abdominal and Inguinal Region.
Description: Log10/cm2 baseline skin flora for abdominal and inguinal regions
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10/cm2 skin flora
Arm/Group | ChloraPrep Hi-Lite Orange - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep Tint 10.5-mL - Abdominal | 3M CHG/IPA Prep Tint 26-mL - Abdominal | ChloraPrep Hi-Lite Orange - Inguinal | Normal Saline - Inguinal | 3M CHG/IPA Prep Tint 10.5-mL - Inguinal | 3M CHG/IPA Prep Tint 26-mL - Inguinal
Number analyzed (Participants) | 198 | 62 | 205 | 201 | 200 | 59 | 204 | 203
log10/cm2 skin flora | 3.31 (0.391) | 3.27 (0.342) | 3.35 (0.427) | 3.31 (0.370) | 5.44 (0.479) | 5.40 (0.448) | 5.44 (0.490) | 5.42 (0.469)

7. Secondary Outcome: Safety as Assessed by Skin Irritation (Dryness, Edema, Erythema, Rash) Rating Score
Description: Skin irritation (dryness, edema, erythema, rash) assessed on the test sites using a 0-3 rating scale: 0=no reaction, 1=mild, 2=moderated, 3=severe
Time Frame: Assessed at baseline (pre-treatment) and 10 minute post-treatment and 6 hour post-treatment.
Population: The primary safety analysis data set used an Intent to Treat population.
Measure: Number; unit: test sites on skin
Arm/Group | ChloraPrep Hi-Lite Orange - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep Tint 10.5-mL - Abdominal | 3M CHG/IPA Prep Tint 26-mL - Abdominal | ChloraPrep Hi-Lite Orange - Inguinal | Normal Saline - Inguinal | 3M CHG/IPA Prep Tint 10.5-mL - Inguinal | 3M CHG/IPA Prep Tint 26-mL - Inguinal
Number analyzed (Participants) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
test sites on skin
  Baseline Dryness-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  Baseline Dryness-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Dryness-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Dryness-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Edema-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  Baseline Edema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Edema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Edema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Erythema-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  Baseline Erythema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Erythema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Erythema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Rash-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  Baseline Rash-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Rash-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Rash-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Dryness-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  10 minute Dryness-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Dryness-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Dryness-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Edema-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  10 minute Edema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Edema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Edema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Erythema-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  10 minute Erythema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Erythema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Erythema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Rash-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  10 minute Rash-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Rash-Mild (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  10 minute Rash-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Dryness-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  6 hour Dryness-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Dryness-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Dryness-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Edema-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  6 hour Edema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Edema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Edema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Erythema-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  6 hour Erythema-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Erythema-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Erythema-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Rash-No Reaction (0) | 247 | 74 | 246 | 245 | 236 | 70 | 238 | 238
  6 hour Rash-Mild (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Rash-Moderate (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  6 hour Rash-Severe (3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected on treatment day. By definition, all AEs were treatment-emergent.
Groups:
- ChloraPrep Hi-Lite Orange - Abdominal: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 26-mL applied topically to the abdominal region for 30 seconds.
  ChloraPrep Hi-Lite Orange: Apply topically.
- ChloraPrep Hi-Lite Orange - Inguinal: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70% 26-mL applied topically to the inguinal region for 2 minutes.
  ChloraPrep Hi-Lite Orange: Apply topically.
Arm/Group | ChloraPrep Hi-Lite Orange - Abdominal | Normal Saline - Abdominal | 3M CHG/IPA Prep Tint 10.5-mL - Abdominal | 3M CHG/IPA Prep Tint 26-mL - Abdominal | ChloraPrep Hi-Lite Orange - Inguinal | Normal Saline - Inguinal | 3M CHG/IPA Prep Tint 10.5-mL - Inguinal | 3M CHG/IPA Prep Tint 26-mL - Inguinal
All-Cause Mortality (participants affected / at risk) | 0/247 | 0/74 | 0/246 | 0/245 | 0/236 | 0/70 | 0/238 | 0/238
Serious Adverse Events (participants affected / at risk) | 0/247 | 0/74 | 0/246 | 0/245 | 0/236 | 0/70 | 0/238 | 0/238
Other Adverse Events (participants affected / at risk) | 0/247 | 0/74 | 0/246 | 0/245 | 0/236 | 0/70 | 0/238 | 0/238

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes